CLINICAL TRIAL: NCT04089345
Title: Stelara fOr ChRonic AntibioTic rEfractory pouchitiS (SOCRATES): A Belgian Open Label Multicenter Pilot-study
Brief Title: Stelara fOr ChRonic AntibioTic rEfractory pouchitiS
Acronym: SOCRATES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNTO1275UCO2001
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2021-04

CONDITIONS: Pouchitis
MeSH Terms: conditions — Pouchitis | interventions — Ustekinumab

STUDY DESIGN:
Intervention Model Description: open label pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Open label ustekinumab (Experimental): All patients will receive intravenously (IV) ustekinumab ~6mg/kg at baseline and subcutaneously (SC) ustekinumab 90mg every 8 weeks thereafter until Week 48. All subjects will receive concomitant antibiotic treatment with ciprofloxacin or metronidazole from baseline through Week 4. Intravenous induction doses will be 260mg for patients <55kg, 390mg for patients between 55 and 85kg, and 520mg for patients with a body weight >85 kg.
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — All patients will receive intravenously (IV) ustekinumab ~6mg/kg at baseline and subcutaneously (SC) ustekinumab 90mg every 8 weeks thereafter until Week 48.
  Other Names: Stelara

SUMMARY:
To evaluate the efficacy and safety of ustekinumab in the treatment of chronic antibiotic refractory and relapsing pouchitis.

DETAILED DESCRIPTION:
This study is a Belgian prospective open label multicenter study to evaluate the efficacy and safety of ustekinumab in the treatment of relapsing or chronic antibiotic refractory pouchitis during a 48-week treatment period. Twenty subjects with a RPC and IPAA for UC who have developed relapsing or chronic antibiotic refractory pouchitis will be enrolled.

All patients will receive intravenously (IV) ustekinumab ~6mg/kg at baseline and subcutaneously (SC) ustekinumab 90mg every 8 weeks thereafter until Week 48. All subjects will receive concomitant antibiotic treatment with ciprofloxacin or metronidazole from baseline through Week 4. Intravenous induction doses will be 260mg for patients <55kg, 390mg for patients between 55 and 85kg, and 520mg for patients with a body weight >85 kg.

Clinical and biochemical evaluation will be planned every 8 weeks. Efficacy will be assessed at Week 16 and Week 48 using mPDAI and PDAI scores, therefor a pouchoscopy with biopsy sampling will be performed. Patients who do not achieve partial response (reduction of mPDAI score by ≥2 points from baseline) at Week 16 will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a history of ileal pouch-anal anastomosis (IPAA) for ulcerative colitis (UC)
* The subject has pouchitis that is (a) relapsing or (b) chronic antibiotic refractory, defined by an mPDAI score ≥5 assessed as the average from 3 days immediately prior to the baseline endoscopy visit and a minimum endoscopic subscore of 2 (outside the staple or suture line) with either (a) ≥3 recurrent episodes within the last year, each treated with ≥2 weeks of antibiotic or other prescription therapy, or (b) requiring maintenance antibiotic therapy taken continuously for ≥4 weeks immediately prior to the baseline endoscopy visit

Exclusion Criteria:

* Crohn's disease (CD), CD-related complications of the pouch (pouch fistula, pouch strictures, ulcerations in the pre-pouch ileum without pouchitis), irritable pouch syndrome (IPS), isolated or predominant cuffitis, infectiouw pouchitis, diverting ostomy or mechanical complications of the pouch
* Previous treatment with an anti-IL12/23 or an anti-IL23 antibody
* Any investigational or approved biologic agent within 30 days of baseline
* Nonbiologic investigational therapy or tofacitinib within 30 days prior to baseline
* Active or untreated latent tuberculosis (TB)
* Chronic hepatitis B virus (HBV) infection, chronic hepatitis C virus (HCV) infection, a known history of human immunodeficiency virus (HIV) infection (or is found to be seropositive at screening) or subject is immunodeficient
* Active severe infection (e.g. sepsis, cytomegalovirus, listeriosis or C. difficile)
* History of malignancy or current malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects achieving clinically relevant steroid-free remission | 16 weeks after baseline
  mPDAI score <5 and a reduction by ≥2 points from baseline

SECONDARY OUTCOMES:
The percentage of subjects achieving clinically relevant steroid-free remission | 48 weeks after baseline
  mPDAI score <5 and a reduction by ≥2 points from baseline, without need for steroids
The percentage of subjects achieving partial response | 16 weeks after baseline
  reduction of mPDAI score by ≥2 points from baseline
The percentage of subjects achieving partial response | 48 weeks after baseline
  reduction of mPDAI score by ≥2 points from baseline
Time to clinically relevant remission | Within 48 weeks after baseline
  Time to mPDAI score <5 and a reduction by ≥2 points from baseline
Change in mPDAI endoscopic subscore | At Week 16 and 48 compared to baseline
  Change in mPDAI endoscopic subscore from baseline
Change in mPDAI symptomatic subscore | At Week 16 and 48 compared to baseline
  Change in mPDAI symptomatic subscore from baseline
Change in total mPDAI score | At Week 16 and 48 compared to baseline
  Change in total mPDAI score from baseline
Change in European Quality of Life 5 Dimensions (EQ-5D) | At Week 16, 32 and 48 compared to baseline
  Change in European Quality of Life 5 Dimensions (EQ-5D) from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, MD, PhD, Principal Investigator — UZ Leuven
Locations (3):
- Belgium (3):
  - UZ Leuven, Leuven, Flanders
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU de Liège, Sart Tilman, Liège

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication

REFERENCES:
- [Derived] Outtier A, Louis E, Dewit O, Reenaers C, Schops G, Lenfant M, Pontus E, De Hertogh G, Verstockt B, Sabino J, Vermeire S, Ferrante M. Efficacy and Safety of Ustekinumab for Chronic Pouchitis: A Prospective Open-label Multicenter Study. Clin Gastroenterol Hepatol. 2024 Dec;22(12):2468-2474.e1. doi: 10.1016/j.cgh.2024.04.030. Epub 2024 May 14. PMID 38750870